CLINICAL TRIAL: NCT06568692
Title: A Phase 2, Open-Label Study of PCS6422 With Capecitabine in Patients With Advanced or Metastatic Breast Cancer
Brief Title: A Phase 2 Study of PCS6422 With Capecitabine in Patients With Advanced or Metastatic Breast Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Processa Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PCS6422-BC-01
Record Dates: First submitted 2024-08-21; First posted 2024-08-23 (Actual); Last update posted 2025-06-19 (Actual); Status verified 2025-06

CONDITIONS: Breast Cancer; TNBC - Triple-Negative Breast Cancer; HER2-negative Breast Cancer
Keywords: HR positive; Advanced Breast Cancer; Metastatic Breast Cancer
MeSH Terms: conditions — Breast Neoplasms; Triple Negative Breast Neoplasms | interventions — Capecitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- PCS6422 40 mg + Capecitabine 300 mg (Experimental): Fixed single dose of PCS6422 administered with Capecitabine 150 mg BID over 7 days
  Interventions: Drug: PCS6422 and capecitabine
- PCS6422 40 mg + Capecitabine 450 mg or 150 mg (Experimental): Fixed single dose of PCS6422 administered with Capecitabine 225 mg or 75 mg BID over 7 days
  Interventions: Drug: PCS6422 and capecitabine
- Capecitabine 2000 mg/m2 (Active Comparator): Standard capecitabine dose at 1000 mg/m2 BID
  Interventions: Drug: Capecitabine

INTERVENTIONS:
Drug: PCS6422 and capecitabine — PCS6422 is an experimental drug that, when combined with capecitabine, may make the immune response more active against cancer.
  Arms: PCS6422 40 mg + Capecitabine 300 mg; PCS6422 40 mg + Capecitabine 450 mg or 150 mg
Drug: Capecitabine — Commercially available capecitabine is a commonly used oral fluoropyrimidine.
  Arms: Capecitabine 2000 mg/m2

SUMMARY:
This is an adaptive Phase 2, open-label, randomized, multi-center study evaluating up to 2 regimens of PCS6422 with capecitabine (Cap) vs. standard dose of Cap alone in patients with advanced or metastatic breast cancer. The goal of the study is to assess the efficacy and safety of PCS6422 + Cap as a treatment option for patients with advanced or metastatic breast cancer who are not eligible for anthracycline- or taxane-containing therapies, or other available therapies, including PD-1 or PARP inhibitors.

DETAILED DESCRIPTION:
This is an adaptive Phase 2, open-label, randomized, multi-center study evaluating up to 2 regimens of PCS6422 with Cap vs. standard dose of Cap alone in patients with advanced or metastatic breast cancer who are not eligible for anthracycline- or taxane-containing therapies, or other available therapies, including PD-1 or PARP inhibitors. The goal of the study is to assess the efficacy and safety of PCS6422 + Cap as a treatment option for patients with advanced or metastatic breast cancer who have been treated with chemotherapy in the metastatic setting.

ELIGIBILITY:
Inclusion Criteria:

1. Aged ≥18 years at Screening
2. Diagnosis of histologically confirmed breast cancer that is unresectable. The following subsets of breast cancer are included:

   1. Patients with triple-negative breast cancer, advanced or metastatic
   2. Patients with hormone receptor (HR) positive, ER positive, HER2 negative advanced or metastatic breast cancer
3. Has measurable disease in accordance with RECIST 1.1 obtained by imaging within 28 days prior to C1D1
4. Other therapies are not indicated (eg, resistant or intolerant to taxanes and/or an anthracycline-containing regimen) for treatment of advanced or metastatic breast cancer
5. Has a life expectance of at least 24 weeks
6. Has Eastern Cooperative Oncology Group Performance Status (ECOG PS) 0 or 1 at screening
7. Has adequate bone marrow, liver, and renal function as assessed by the following laboratory requirements conducted within 7 days before C1D1 (Note: labs will also be repeated pre-dose on C1D1 to confirm eligibility): a. Hemoglobin ≥9 g/dL (≥90 g/L) b. Adequate renal function by estimated glomerular filtration rate (eGFR) defined as a creatinine clearance >50 mL/min (>0.84 mL/s) (Cockcroft-Gault equation) and normalized to body surface area c. Peripheral absolute neutrophil count (ANC) of ≥1.5×109/L d. Platelet count of ≥100×109/L without growth factor/transfusion e. Total bilirubin <1.5× upper limit of normal (ULN); or ≤3×ULN if the patient has Gilbert's disease f. Aspartate aminotransferase (AST) or alanine aminotransferase (ALT) <2.5×ULN, with liver metastasis <5×ULN g. International normalized ratio (INR) <1.5 and prothrombin time (PT) ≤1.5×ULN, unless both of the following conditions are met: i. Patient is receiving anticoagulant therapy, and ii. PT or partial thromboplastin time (PTT) is within therapeutic range of intended use of anticoagulant h. Activated partial thromboplastin time (aPTT) ≤1.5×ULN, unless both of the following conditions are met: i. Patient is receiving anticoagulant therapy, and ii. PT or PTT is within therapeutic range of intended use of anticoagulants

Exclusion Criteria:

1. Received any line of treatment for advanced or metastatic breast cancer within 21 days or 5 half-lives (whichever is longer) prior to randomization
2. Currently receiving any hormone replacement therapy, unless discontinued within 21 days prior to randomization
3. Received IV 5-FU or oral 5-FU analog in the 4 weeks prior to C1D1
4. Received DPD inhibitor within 4 weeks prior to C1D1
5. Has homozygous or compound heterozygous DPYD variants that result in complete or near-complete absence of DPD activity
6. Cardiac:

   1. Has history or presence of clinically significant abnormal 12-lead electrocardiogram (ECG) results, in the Medical Monitor or Investigator's opinion
   2. Has prolonged QTc (with Fridericia's correction) of >480 msec performed at Screening
   3. Has a history of prolonged QTc interval, ventricular tachycardia/fibrillation or significant ventricular arrhythmia, or Torsades de Pointes, or a history of ventricular ablation for arrhythmia
   4. Has congenital long QT syndrome or a family history of long QT syndrome
   5. Has other clinically significant cardiac disease including, but not limited to, myocardial infarction, unstable angina, cardiac or other vascular stenting, angioplasty, or surgery ≤12 months prior to randomization, congestive heart failure

      * Class II per the New York Heart Association, or history of myocarditis
7. Is pregnant or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2024-10-02 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Evaluation of Objective Response Rate (ORR) | Up to 24 weeks post End of Treatment (EoT)
  The proportion of patients who achieved a confirmed complete response (CR) or partial response (PR) according to Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST 1.1)
Number of patients with adverse events (AEs) | During treatment, an average of 8 months
  Frequency, duration, and severity of AEs across treatment groups

SECONDARY OUTCOMES:
Evaluation of Disease Control Rate (DCR) | Up to 24 weeks post End of Treatment (EoT)
  The proportion of patients with objective evidence of CR or PR or stable disease (SD) according to RECIST 1.1
Evaluation of Duration of Response (DOR) | Up to 24 weeks post End of Treatment (EoT)
Evaluation of Time to Response (TTR) | Every 12 weeks during treatment
Evaluation of Progression Free Survival (PFS) | Up to 24 weeks post End of Treatment (EoT)

CONTACTS AND LOCATIONS:
Locations (13):
- United States (13):
  - Arizona Oncology Associates, Tucson, Arizona
  - Valkyrie Clinical Trials, Los Angeles, California
  - FOMAT Medical Research, Oxnard, California
  - AP Medical Research, Miami, Florida
  - Moffitt Cancer Center, Tampa, Florida
  - Northwest Cancer Center, Dyer, Indiana
  - University of Maryland Medical Center (UMMC), Baltimore, Maryland
  - Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey
  - Clinical Research Alliance, Westbury, New York
  - Gabrail Cancer Center Research, Canton, Ohio
  - SCRI Oncology Partners, Nashville, Tennessee
  - Texas Oncology PA (Austin), Austin, Texas
  - Texas Oncology PA (San Antonio), San Antonio, Texas